CLINICAL TRIAL: NCT02685969
Title: Characterization of Cerebral Amyloid Deposition With 18F-Flutemetamol PET and of Glucose Metabolism With 18F-FDG PET in Individuals Enrolled in the ALFA Project.
Brief Title: Brain Characterization of Amyloid Protein and Glucose Metabolism of ALFA Project Participants
Status: Recruiting | Type: Observational
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Collaborators: Hospital Clinic of Barcelona (Other); General Electric (Industry)
Responsible Party: Sponsor
Other Study IDs: PET FLUTEMETAMOL-FDG/BBRC2015
Record Dates: First submitted 2016-02-15; First posted 2016-02-19 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer's Disease
Keywords: Prevention; Positron Emission Tomography
MeSH Terms: conditions — Alzheimer Disease | interventions — flutemetamol; Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 18F-Flutemetamol & 18F-FDG PET scans: All study participants will be assessed by PET scan with 18F-Flutemetamol & 18F-FDG PET scans.
  Interventions: Procedure: 18F-Flutemetamol & 18F-FDG

INTERVENTIONS:
Procedure: 18F-Flutemetamol & 18F-FDG — Characterization of cerebral amyloid deposition with 18F-Flutemetamol PET and glucose metabolism 18F-FDG PET.

SUMMARY:
Study to understand factors related with the preclinical stages of Alzheimer's Disease and investigate markers that predict its progression.

Cross-sectional and single arm study performed on a subgroup of individuals recruited in the ALFA project.

Study without therapeutic interest for the research participants (440 participants of the ALFA project who have been selected for being cognitively healthy and in their vast majority are direct descendants of patients diagnosed with Alzheimer's Disease).

Each study candidate will be selected from the ALFA project (STUDY 45-65 FPM/2012) according to their clinical characteristics, their compliance to selection criteria and their desire to participate in this study.

After signing this study's specific informed consent form, the neuropsychological screening and the brain MRI acquisition will be performed. Once all inclusion criteria are checked, the PET scans with 18F-Flutemetamol and 18F-FDG will be performed

DETAILED DESCRIPTION:
18F-Flutemetamol scans will be categorized as either positive or negative according to the standardized uptake value ratio (a quantitative measurement based on a ratio of mean target cortex activity divided by that in a cerebellar reference region). Participants with a SUVr over 1.56 will be classified as positive and, otherwise, as negative.

ELIGIBILITY:
Inclusion Criteria:

* To sign the study informed consent form approved by the corresponding authorities.
* Men and women enrolled in the ALFA project (STUDY 45-65 FPM/2012).
* Participants with a cerebral MRI (magnetic resonance imaging) not suggestive of radiological incidental findings constituting an exclusion criterion.
* Cognition within psychometrically normal ranges: MMSE (Mini Mental State Examination ≥26 and Semantic Fluency (animals) ≥12.
* Score of 0 in the CDR scale (Clinical Dementia Rating).
* Good knowledge of the language and being literate.
* Female participants should be post-menopausal or present a negative pregnancy test at the moment of PET acquisition.

Exclusion Criteria:

* Present cognitive impairment.
* Presence of clinically relevant psychiatric disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV-TR) criteria: major depressive disorder, generalized anxiety disorder, schizophrenia or bipolar disorder.
* Individuals with visual and/or hearing impairment.
* History of encephalitis, ictus or seizures excluding feverish convulsions during childhood.
* Severe cerebral macrovascular (i.e., multi-stroke) disease or brain tumor (metastasis/brain cancer) as verified by magnetic resonance imaging (MRI).
* Any contraindication to MRI acquisition, (i.e., metal implants) or phobia to performing the scan as determined by the onsite physician.
* Previous participation in a clinical study involving an investigational pharmaceutical product within 30 days prior to screening and/or administration of a radiopharmaceutical within 10 radioactive half-lives prior to study drug administration in this study.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 440 participants enrolled in the ALFA project (STUDY 45-65 FPM/2012) will be selected and physiologically characterized with 18F-Flutemetamol and 18F-FDG PET scans.
Sampling Method: Non-Probability Sample
Enrollment: 570 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of a positive 18F-Flutemetamol scan | Baseline
  To study the prevalence of a positive 18F-Flutemetamol PET scan in a cohort of cognitively healthy, at-risk of developing AD participants.

SECONDARY OUTCOMES:
Prevalence of the different stages of preclinical AD according to the NIA-AA criteria | Baseline
  Analysis of amiloid PET acquired

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Molinuevo, MD, PhD, Principal Investigator — Scientific Director
Locations (1):
- BarcelonaBeta Brain Research Center, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brugulat-Serrat A, Sanchez-Benavides G, Cacciaglia R, Salvado G, Shekari M, Collij LE, Buckley C, van Berckel BNM, Perissinotti A, Ninerola-Baizan A, Mila-Aloma M, Vilor-Tejedor N, Operto G, Falcon C, Grau-Rivera O, Arenaza-Urquijo EM, Minguillon C, Fauria K, Molinuevo JL, Suarez-Calvet M, Gispert JD; ALFA Study. APOE-epsilon4 modulates the association between regional amyloid deposition and cognitive performance in cognitively unimpaired middle-aged individuals. EJNMMI Res. 2023 Mar 1;13(1):18. doi: 10.1186/s13550-023-00967-6. PMID 36856866
- [Derived] Grau-Rivera O, Navalpotro-Gomez I, Sanchez-Benavides G, Suarez-Calvet M, Mila-Aloma M, Arenaza-Urquijo EM, Salvado G, Sala-Vila A, Shekari M, Gonzalez-de-Echavarri JM, Minguillon C, Ninerola-Baizan A, Perissinotti A, Simon M, Kollmorgen G, Zetterberg H, Blennow K, Gispert JD, Molinuevo JL; ALFA Study. Association of weight change with cerebrospinal fluid biomarkers and amyloid positron emission tomography in preclinical Alzheimer's disease. Alzheimers Res Ther. 2021 Feb 17;13(1):46. doi: 10.1186/s13195-021-00781-z. PMID 33597012
- [Derived] Salvado G, Molinuevo JL, Brugulat-Serrat A, Falcon C, Grau-Rivera O, Suarez-Calvet M, Pavia J, Ninerola-Baizan A, Perissinotti A, Lomena F, Minguillon C, Fauria K, Zetterberg H, Blennow K, Gispert JD; Alzheimer's Disease Neuroimaging Initiative, for the ALFA Study. Centiloid cut-off values for optimal agreement between PET and CSF core AD biomarkers. Alzheimers Res Ther. 2019 Mar 21;11(1):27. doi: 10.1186/s13195-019-0478-z. PMID 30902090